CLINICAL TRIAL: NCT05042609
Title: A Phase 3 Randomized, Active-Controlled, Double-Masked Study to Evaluate the Safety and Efficacy of TRS01 Eye Drops in the Treatment of Subjects With Active Non-infectious Anterior Uveitis Including Subjects With Uveitic Glaucoma
Brief Title: A Study of TRS01 in Subjects With Active Non-infectious Anterior Uveitis Including Subjects With Uveitic Glaucoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tarsier Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRS4Vision
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Non-infectious Anterior Uveitis; Uveitic Glaucoma
MeSH Terms: interventions — Masks

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRS01 (Experimental)
  Interventions: Drug: TRS01
- Active comparator (Active Comparator)
  Interventions: Drug: FDA approved steroid eye drop (masked)

INTERVENTIONS:
Drug: TRS01 — TRS01 eye drops Dosed four times a day (QID)
  Arms: TRS01
Drug: FDA approved steroid eye drop (masked) — FDA approved steroid eye drop Dosed four times a day (QID)
  Arms: Active comparator

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of TRS01 eye drops compared to active comparator in subjects with active non-infectious anterior uveitis with or without uveitic glaucoma

ELIGIBILITY:
Inclusion Criteria:

* At sites in the US: Male or female up to and including 75 years of age (including all pediatric age groups). At sites in the Europe: Male or female between 18 and 70 years of age, inclusive.
* Diagnosed with active non-infectious anterior uveitis with anterior chamber cell Grade 2 (6-15 cells) or Grade 3 (16-30 cells) in the study eye that are without any treatment or with Stable Medical Therapy requiring further treatment.
* Have Best Corrected Visual Acuity (BCVA) vision ≥ 65 letters in the non-study eye using Early Treatment Diabetic Retinopathy Study (ETDRS).

Exclusion Criteria:

* Pregnant or breastfeeding females or females.
* History of or active significant ocular disease in either eye.
* Uncontrolled intraocular pressure (IOP; defined as >27mmHg) or narrow angle glaucoma in either eye and/or are at risk of angle closure with dilating.
* Poor posterior view due to limitation of dilation or media opacity that limits ability to examine the posterior segment.
* Cancer or melanoma that is actively treated with immunotherapy.
* Certain clinically significant systemic diseases or conditions.
* Receiving specific medication/interventions as specified per protocol.

Ages: 0 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Anterior Chamber Cell (ACC) grade on Day 28 | 28 days
  For FDA submission: the proportion of subjects with Anterior Chamber Cell (ACC) Grade=0 (0 cells) on Day 28 in the study eye.
  For submission to European Medicines Agency (EMA) related countries: the proportion of subjects with ACC Grade = 0 or 1 on Day 28 in the study eye.

SECONDARY OUTCOMES:
Change from baseline (Day 1) in ACC Grade on Day 28 in the study eye | 28 days
Anterior Chamber Cell (ACC) grade on Day 21 | 21 days
  For FDA submission: Proportion of subjects with ACC Grade=0 on Day 21 in the study eye.
  For submission to EMA related countries: Proportions of subjects with ACC Grade = 0 or 1 on Day 21 in the study eye.
Change from baseline in ACC Grade on Day 21. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Lexitas Clinical Trials, Study Director — Lexitas
Locations (29):
- United States (19):
  - La Jolla, La Jolla, California
  - Los Angeles, Los Angeles, California
  - Los Angeles 2, Los Angeles, California
  - Aurora, Aurora, Colorado
  - Lakewood, Lakewood, Colorado
  - Jacksonville, Jacksonville, Florida
  - Winter Haven, Winter Haven, Florida
  - Marietta, Marietta, Georgia
  - Boston, Boston, Massachusetts
  - Waltham, Waltham, Massachusetts
  - Washington, MO, Washington, Missouri
  - Palisades Park, Palisades Park, New Jersey
  - Winston-Salem, Winston-Salem, North Carolina
  - Nashville, Nashville, Tennessee
  - Austin, Austin, Texas
  - Plano, Plano, Texas
  - San Antonio 2, San Antonio, Texas
  - San Antonio, San Antonio, Texas
  - Norfolk, Norfolk, Virginia
- France (4):
  - Dijon, Dijon
  - Lyon, Lyon
  - Nantes, Nantes
  - Paris, Paris
- Germany (6):
  - Bonn, Bonn
  - Düsseldorf, Düsseldorf
  - Freiburg, Freiburg im Breisgau
  - München, München
  - Munster, Münster
  - Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No